CLINICAL TRIAL: NCT01365910
Title: An Investigator Initiated, Phase II Study of Linifanib in Patients With Advanced, Refractory Colorectal Cancer Expressing Mutated kRas
Brief Title: Linifanib in Treating Patients With Advanced, Refractory Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis determined the study did not meet criteria to proceed
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Jordan Berlin, MD, Professor of Medicine; Clinical Director, GI Oncology Program; Director, Phase I Program; Medical Director, Clinical Trials Shared Resources; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC GI 1058; NCI-2011-00833 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Results first posted 2014-08-26 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — linifanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (enzyme inhibitor) (Experimental): Patients receive linifanib PO QD. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: linifanib

INTERVENTIONS:
Drug: linifanib — Given PO
  Other Names: ABT-869; multitargeted receptor tyrosine kinase inhibitor ABT-869

SUMMARY:
This phase II trial studies how well Linifanib works in treating patients with advanced, refractory colorectal cancer expressing k-Ras mutations. Linifanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To achieve an overall response rate of 15% or more.

SECONDARY OBJECTIVES:

I. Determine progression free survival. II. Determine overall survival. III. Evaluate toxicity profile of ABT 869 (linifanib) in this patient population.

OUTLINE:

Patients receive Linifanib orally (PO) once daily (QD). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 2 years, and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal cancer refractory to at least 1 but no more than 3 systemic chemotherapy regimens
* Patients must have received one standard chemotherapy regimen in the metastatic setting
* Established Ras-mutant tumor status (archived specimens are okay and this test can have been performed at local laboratories)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* The subject must have adequate bone marrow and organ function, defined as follows:
* Hemoglobin ≥ 9g/dL
* Platelets >100,000,
* Absolute neutrophil count (ANC) > 1000/uL,
* Serum creatinine < 1.5 x upper limit of normal,
* Total bilirubin < 1.5 x the upper limit of normal,
* AST and ALT ≤ 2.0 x upper limit of normal (or ≤ 5 x ULN in the presence of liver metastases)
* Measurable disease, defined as at least 1 unidimensionally measurable lesion on a computed tomography (CT) scan or magnetic resonance imaging (MRI) as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 7 days of study treatment; surgically sterile and/or postmenopausal women must be amenorrheic for at least 12 months to be considered of non-child-bearing potential
* Female subjects of child-bearing potential and male subjects must agree to use adequate contraception prior to study entry, for the duration of study participation and up to two months after the last dose of ABT 869; adequate contraception methods should be used consistently and correctly and include the following:
* Total abstinence from sexual intercourse (minimum one complete menstrual cycle)
* A vasectomized partner
* Hormonal contraceptives (oral, parenteral or transdermal) for at least 3 months prior to study drug administration
* Double-barrier method (condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or cream)
* The subject must be willing and able to comply with the protocol for the duration of the study, including undergoing treatment and scheduled visits and examinations
* The subject must have given written informed consent prior to the initiation of any screening or study-specific procedures
* Ability to understand and the willingness to sign a written informed consent; a signed informed consent must be obtained prior to any study-specific procedures
* Patients must be at least 14 days status post last day of prior chemotherapy (at least 28 days since last dose of bevacizumab) and have recovered to grade =< 1 from all chemotherapy-associated side effects
* Patients must have the ability to swallow pills

Exclusion Criteria:

* Untreated central nervous system (CNS) metastases; patients may have CNS metastases from any timeframe as long as they are treated and not progressing; brain imaging is not required if there is no clinical suspicion of brain metastases
* Pregnant or lactating females are excluded
* Uncontrolled hypertension defined as systolic blood pressure (BP) > 140 and/or diastolic BP > 90 initially evaluated on day of study eligibility determination (when laboratory parameters are assessed), but must be maintained on day of study initiation; (If a patient is found to have a value outside the range above, repeat BP may be assessed and if at subsequent readings x 2 (taken in clinic at least 15 minutes apart) criteria are met, the patient can then be eligible; initiation or modification of antihypertensives is allowed to achieve adequate BP for eligibility; finally, in the case that subsequent determinations are required, the BP assessment that counts towards eligibility is the reading on the day of study initiation); (note: a clinic BP reading without the patient having been at rest for 15 minutes or with the wrong cuff size can be repeated the same day for eligibility criteria to be determined
* Active bleeding or history of bleeding from cancer related events
* History of cerebral vascular accident (CVA) or transient ischemic attack (TIA) or recent myocardial infarction (MI) (< 6 months)
* Active ulcerative colitis, Crohn's disease or Celiac disease that could interfere with the absorption of the drug
* Current use of therapeutic anticoagulation; low dose anticoagulation for catheter prophylaxis is permitted; Lovenox is permitted for prophylaxis; (Note: patients who develop thrombosis and are placed on anticoagulation while on this trial may continue on study at the discretion of the investigator)
* The subject has had major surgery within 28 days of Study Day 1
* The subject has had radiation therapy within 14 days of Study Day 1
* The subject had prior bevacizumab within 28 days of study day 1
* No prior treatment with vascular endothelial growth factor (VEGF) receptor tyrosine kinase inhibitors; prior treatment with other investigational agents is allowed
* The subject has a medical condition, which in the opinion of the study investigator, places them at unacceptably high risk for toxicities
* Other active malignancy for which the patient has been treated within the past one year
* Subjects with known human immunodeficiency virus (HIV) infection are excluded
* Subject has documented left ventricular ejection fraction (LVEF) < 50%
* Subject has Proteinuria > grade 1 at baseline measured by urine dipstick (2+ or greater) and confirmed by 24 hour (hr) urine collection (> = 1g/24hrs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Berlin, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (2):
- United States (2):
  - Vanderbilt Cool Springs, Franklin, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clnical Trial — http://www.vicc.org/ct/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study opened June 3, 2011 and continued until June 3, 2013. Patients were enrolled at Vanderbilt-Ingram Cancer Center.
Pre-assignment Details: Thirty-five patients consented to be on this study. Four patients were considered ineligible, and 1 patient withdrew prior to treatment.
Groups:
- Treatment (Enzyme Inhibitor): ABT-869/Linifanib will be administered orally on a daily basis at 17.5 mg/day (fixed dose). The drug is provided in tablets of 2.5 mg or 10 mg tablets.This course of treatment repeats every 28 days until disease progression, intolerability, investigator decision or patient withdrawal of consent.
Period: Overall Study
Arm/Group | Treatment (Enzyme Inhibitor)
Started | 30
Completed | 0
Not Completed | 30
Not completed — Withdrawal by Subject | 7
Not completed — disease progression | 18
Not completed — Adverse Event | 3
Not completed — other complicating disease | 1
Not completed — pt did not get tx, nausea/vomiting | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Enzyme Inhibitor)
Number analyzed (Participants) | 30
Age, Customized [Number; unit: participants]
  Age 20-29 | 1
  Age 40-49 | 4
  Age 50-59 | 10
  Age 60-69 | 10
  Age 70-79 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 24
  More than one race | 2
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Complete Response + Partial Response) With a Target of at Least 15%
Description: Per Response Evaluation in Solid Tumors (RECIST) criteria v. 1.1: measurable lesions: complete response (CR) disappearance of target lesions, partial response (PR) > 30% decrease in the sum of the longest diameter (LD) of target lesions, progressive disease (PD) > 20% increase in the sum of the LD of target lesions or appearance of new lesions, stable disease (SD) neither sufficient decrease nor increase of the sum of smallest sum of the LD of target lesions. Defined as the CR + PR recorded from the start of the treatment until disease progression/recurrence, the exact two-sided 95% confidence intervals will be reported.
Time Frame: Baseline and every 8 weeks, up to 2 years
Population: All patients are included in the analysis on intention-to-treat basis. Analysis is by Kaplan-Meier method, where death is an event, with censoring for non-expired patients at greater of off-study date or last known alive date.
Measure: Median (95% Confidence Interval); unit: percentage of target lesions
Arm/Group | Treatment (Enzyme Inhibitor)
Number analyzed (Participants) | 23
percentage of target lesions | 0 [0 to 0.148]

2. Secondary Outcome: Progression-free Survival
Description: Estimated probable duration of life without disease progression, from on-study date to earlier of progression date or date of death from any cause, using the Kaplan-Meier method with censoring. Disease progression is defined under RECIST v1.1 as >=20% increase in sum of longest diameters of target lesions, unequivocal progression of non-target lesions, or appearance of new lesions.
Time Frame: Every 3 months, up to 2 years
Population: All patients are included in the analysis on intention-to-treat basis. Analysis is by Kaplan-Meier method, where either death or progression is an event, with censoring for non-progressed, non-expired patients at greater of off-study date or last known alive date.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment (Enzyme Inhibitor)
Number analyzed (Participants) | 29
days | 155 [112 to 290]

3. Secondary Outcome: Overall Survival
Description: Estimated probable duration of life from on-study date to date of death from any cause, using the Kaplan-Meier method with censoring.
Time Frame: Every 3 months, up to 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment (Enzyme Inhibitor)
Number analyzed (Participants) | 29
days | 290 [158 to 367]

4. Secondary Outcome: Number of Patients With Each Worst-Grade Toxicity
Description: Count of patients according to the worst-grade toxicity experienced by each, where worst-grade toxicity is per NCI common toxicity criteria: grade 1= mild; grade 2 = moderate; grade 3 = severe; grade 4 = life-threatening; grade 5 = death
  Assessed: days 1 &15 of cycle 1; day 1 of each subsequent 28-day cycle; at 30-day follow-up for two years
Time Frame: date on-study up to 2 years following final dose of study
Population: Total number of patients reported with any toxicity
Measure: Number; unit: participants
Arm/Group | Treatment (Enzyme Inhibitor)
Number analyzed (Participants) | 29
participants
  worst grade toxicity 1 | 0
  worst grade toxicity 2 | 4
  worst grade toxicity 3 | 23
  worst grade toxicity 4 | 1
  worst grade toxicity 5 | 1

ADVERSE EVENTS:
Arm/Group | Treatment (Enzyme Inhibitor)
Serious Adverse Events (participants affected / at risk) | 16/30
Other Adverse Events (participants affected / at risk) | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor) (N=30)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
colonic obstruction (Gastrointestinal disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 2 (2)
ileal perforation (Gastrointestinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (4)
gastric obstruction (Gastrointestinal disorders) | 1 (1)
small intestine obstruction (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
General disorders and administration site conditions Pain (General disorders) | 3 (3)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
dehydration (Metabolism and nutrition disorders) | 3 (3)
confusion (Psychiatric disorders) | 1 (1)
acute kidney injury (Renal and urinary disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor) (N=30)
diarrhea (Gastrointestinal disorders) | 17 (29)
abdominal pain (Gastrointestinal disorders) | 15 (27)
nausea (Gastrointestinal disorders) | 15 (26)
oral pain (Gastrointestinal disorders) | 10 (24)
vomiting (Gastrointestinal disorders) | 10 (16)
mucositis oral (Gastrointestinal disorders) | 7 (10)
constipation (Gastrointestinal disorders) | 6 (9)
dyspepsia (Gastrointestinal disorders) | 5 (5)
hemorrhoids (Gastrointestinal disorders) | 4 (4)
gastrointestinal disorders, other (Gastrointestinal disorders) | 3 (3)
gingival pain (Gastrointestinal disorders) | 2 (2)
fatigue (General disorders) | 24 (78)
pain (General disorders) | 8 (12)
edema (General disorders) | 4 (5)
chills (General disorders) | 2 (2)
fever (General disorders) | 2 (2)
alkaline phosphatase increased (Investigations) | 15 (26)
aspartate aminotransferase increased (Investigations) | 15 (30)
activated partial thromboplastin time increase (Investigations) | 12 (19)
rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
weight loss (Investigations) | 11 (17)
alanine aminotransferase (Investigations) | 9 (15)
platelet count decreased (Investigations) | 8 (16)
white blood cell decreased (Investigations) | 7 (14)
lymphocyte count decreased (Investigations) | 6 (17)
blood bilirubin increased (Investigations) | 4 (9)
neutrophil count decreased (Investigations) | 2 (2)
anexoria (Metabolism and nutrition disorders) | 14 (20)
hyponatremia (Metabolism and nutrition disorders) | 14 (33)
hypoalbuminemia (Metabolism and nutrition disorders) | 13 (20)
hyperglycemia (Metabolism and nutrition disorders) | 7 (11)
hypokalemia (Metabolism and nutrition disorders) | 7 (11)
hypophosphatemia (Metabolism and nutrition disorders) | 7 (9)
hypercalcemia (Metabolism and nutrition disorders) | 3 (3)
dehydration (Metabolism and nutrition disorders) | 2 (2)
hypocalcemia (Metabolism and nutrition disorders) | 2 (3)
hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
proteinuria (Renal and urinary disorders) | 18 (44)
hematuria (Renal and urinary disorders) | 10 (13)
urinary tract obstruction (Renal and urinary disorders) | 2 (2)
hypertension (Vascular disorders) | 20 (109)
hypotension (Vascular disorders) | 3 (3)
anemia (Blood and lymphatic system disorders) | 20 (39)
hoarseness (Respiratory, thoracic and mediastinal disorders) | 12 (14)
cough (Respiratory, thoracic and mediastinal disorders) | 6 (8)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 3 (4)
sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (3)
endrocrine disorders, other (Endocrine disorders) | 8 (13)
hypothyroidism (Endocrine disorders) | 8 (11)
headache (Nervous system disorders) | 7 (10)
dysgeusia (Nervous system disorders) | 6 (8)
dizziness (Nervous system disorders) | 3 (3)
somnolence (Nervous system disorders) | 3 (4)
tremor (Nervous system disorders) | 3 (3)
dysarthria (Nervous system disorders) | 2 (2)
peripheral sensory neuropathy (Nervous system disorders) | 2 (3)
palmar-olantar erthrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 9 (63)
skin and subcutaneous tissue disorders, other (Skin and subcutaneous tissue disorders) | 6 (15)
dry skin (Skin and subcutaneous tissue disorders) | 5 (5)
upper respiratory infection (Infections and infestations) | 3 (3)
urinary tract infection (Infections and infestations) | 3 (4)
arthralgia (Musculoskeletal and connective tissue disorders) | 6 (14)
back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
myalgia (Musculoskeletal and connective tissue disorders) | 3 (4)
extremity pain (Musculoskeletal and connective tissue disorders) | 2 (2)
anxiety (Psychiatric disorders) | 4 (4)
depression (Psychiatric disorders) | 3 (4)
confusion (Psychiatric disorders) | 2 (2)
sinus tachycardia (Cardiac disorders) | 4 (4)
bruising (Injury, poisoning and procedural complications) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes